CLINICAL TRIAL: NCT03684681
Title: The Navigator Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Navigator
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-06

CONDITIONS: Opioid Use; Opioid Dependence; Opioid Abuse; Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Social Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Navigator (Other): Current standard of care
  Interventions: Behavioral: Peer Navigator Intervention
- Social Worker (Other): Current standard of care
  Interventions: Behavioral: Social Work Intervention

INTERVENTIONS:
Behavioral: Peer Navigator Intervention — A peer navigator delivers an intervention to current drug users and uses their own training and real- life experiences to help people meet their goals.
  Arms: Peer Navigator
Behavioral: Social Work Intervention — A hospital social workers uses their own previous training to help people meet their goals.
  Arms: Social Worker

SUMMARY:
In this study, the investigators will investigate if there is a better intervention for patients who present to the emergency department with an overdose or with symptoms consistent with drug use. There are currently two interventions that are routinely used when a patient comes to the Emergency Department with these criteria, and the investigators will compare the two. The first is when hospital social workers uses their own previous training to help people meet their goals. The second is when a person called a peer navigator, who is someone that has been in long-term drug recovery for over two years and has completed a lot of training to work with current drug users, delivers an intervention to current drug users and uses their own training and real- life experiences to help people meet their goals. The investigators hope to determine if patients have better outcomes if they work with one of these two groups.

If a patient agrees to be in the study, the research staff will randomize them (like flipping a coin) to see if they will work with a social worker or a peer navigator. The research staff will distribute a survey in RedCap and the following information will be collected: age, sex, race, type of opioid used, and history of chronic pain, depression or post-traumatic stress disorder. Once the patient is assigned to a group, they will work with their assigned interventionist for the duration of the study. After this, the research team will track the patient to see if they joined an addiction-treatment program within 30 days of when the joined the study. The study team will also track patients to see if they had additional emergency department visits, additional overdoses, and if they successfully completed a treatment program over an 18-month period.

650 patients will be enrolled into the study.

DETAILED DESCRIPTION:
Opioid overdoses are a leading cause of death for Americans under 50 years old, with recent years recording the most opioid overdose deaths on record. US Emergency Departments (EDs) have seen a parallel increase in opioid-related visits (a 100% increase from 2005 - 2014). ED patients presenting for an overdose are at greatly elevated risk for a repeat overdose and death. Thus, an overdose-related ED visit is both a critical and opportune time to prevent recurrent opioid overdose and overdose death through increased uptake in addiction treatment. The most effective means to promote engagement in treatment following an ED visit for opioid overdose remains unknown. To address this critical evidence gap, the investigators will compare the effectiveness of two ED-based behavioral interventions to increase treatment uptake and reduce the risk of future overdose among ED patients who are at greatest risk of accidental drug-related death.

In response to RI's overdose crisis, in 2014, the state's largest ED (Rhode Island Hospital) began a proactive campaign to improve the care of overdose patients. The program includes an ED-based behavioral intervention either by in-house clinical social work staff or peer recovery support specialists ("peer navigators"). Following the introduction of these interventions in the ED, there was 10-fold increase in the proportion of patients engaging in addiction treatment within 30 days of the initial ED visit. While this preliminary data is promising, the effectiveness of the peer navigators versus the social work intervention is not known.

The investigators propose a randomized controlled trial of early ED behavioral interventions following an opioid overdose. The investigators hypothesize that peer navigation will result in greater early treatment engagement and reduction in recurrent opioid overdose compared to a standard intervention delivered by a clinical social worker.

The investigators will determine the effectiveness of peer navigation versus a standard behavioral intervention delivered in the ED to overdose patients and those at risk of recurrent opioid overdose. A total of 650 ED patients will be recruited (n=325 per arm) and followed for 18 months. Effectiveness will be measured objectively through linkage to administrative statewide databases, with two primary endpoints: (1) engagement in formal addiction treatment (e.g., inpatient services, outpatient services, medication assisted treatment (MAT)) from a licensed substance abuse treatment provider within 30 days following the ED visit, and (2) reduction in 18-month recurrent ED visits for an opioid overdose. Exploratory outcomes of interest are: overdose fatality, repeat ED visits related to opioids, and successful completion of an addiction treatment program and/or long-term retention in MAT.

The investigators will explore if there is heterogeneity of treatment effect related to patient characteristics. The investigators anticipate that there will be individuals within each treatment arm who will vary in their response to the intervention. Specifically, the investigators will examine if the effects of the interventions are modified by baseline characteristics such as age, sex, race, type of opioid used, and history of comorbid chronic pain, depression or PTSD. Understanding these factors will allow us to further optimize subsequent interventions.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18 years of age or older
* Treatment for an opioid overdose or identified as having had an opioid overdose in the past 12 months or are being treated for a visit related to illicit opioid use (e.g., abscess, opioid withdrawal)
* Able to provide informed consent.

Exclusion Criteria:

* Less than 18 years of age
* Previously enrolled in the study
* In police custody
* Incarcerated
* Live outside of Rhode Island
* Pregnant
* Critically ill or injured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who are admitted to a formal addiction treatment program within thirty days following the initial ED visit. | 30 days
  Engagement in addiction treatment will be defined as the proportion who are admitted to a formal addiction treatment program within thirty days following the initial ED visit. The research team will be using BHDDH and Prescription Drug Monitoring Program (PDMP) records. The BHDDH database contains information on all admissions to publicly funded substance abuse treatment programs in the state. The RI PDMP manages a database that contains information on all prescriptions for schedule II-IV substances filled in the state. The database is updated daily; all pharmacies are required to report prescriptions within 48-hours of the fill date. All records will be linked deterministically to participant data using identifiable information (e.g., name, social security number) within the Stronghold computing environment, a HIPAA-compliant server maintained by the team at Brown University.
The proportion of participants who are treated in any Rhode Island ED for an opioid overdose at any time during the 18-month follow-up period following the initial ED visit. | 18 months
  The proportion of participants who are treated in any Rhode Island ED for an opioid overdose at any time during the 18-month follow-up period following the initial ED visit, will be assessed by first accessing the electronic medical records (EMRs) of the 12 EDs in Rhode Island (RI) through the Rhode Island Quality Institute Statewide Health Information Exchange. This unified data system provides access to EMR data from all major health systems in RI, capturing repeat visits for an opioid overdose that occur in all 12 EDs in RI. Secondly the research team will query the RI Department of Health (RIDOH) Opioid 48-Hour Overdose Surveillance System which mandates all suspected opioid overdose cases presenting to an RI hospital be reported to the department within 48 hours. This data source will capture recurrent overdoses not identified by ICD codes in the unified EMR data system, and also contains additional fields of interest (e.g., pre-existing risk factors for overdose).

SECONDARY OUTCOMES:
Compare the the time to subsequent opioid overdose rates between groups. | 18 month
  The principal investigator will use Breslow's method to test if the time to subsequent opioid overdose rates differs between the groups.
Successful completion or retention in addiction treatment | 18 month
  Successful completion and/or retention in addiction treatment will be defined based on discharge data collected in BHOLD and prescription refill data in the PDMP. The principal investigator will examine the time to ED visit for an opioid overdose using a Kaplan-Meier analysis. Patients will be censored at the end of the 18-month follow-up period, considered the last point of contact.
Overdose death | 18 months
  Cox proportional hazards modeling will be used to estimate hazard ratios (HRs) and corresponding 95% confidence intervals (CIs) for occurrence of repeat overdose between groups. HRs will be adjusted for clinical and demographic characteristics believed to predict the outcome of opioid overdose in order to adjust for possible residual confounding and treatment-factor interactions.
Heterogeneity of intervention effect | 18 months
  The principal investigator will perform stratified subgroup analyses to determine if treatment effects vary between groups of individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Beaudoin, MD, Principal Investigator — Brown Emergency Medicine
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Chambers LC, Li Y, Hallowell BD, Langdon KJ, Samuels EA, Mahoney LA, Beaudoin FL, Marshall BDL. Effect of a peer-led emergency department behavioral intervention on non-fatal opioid overdose: 18-month outcome in the Navigator randomized controlled trial. Addiction. 2024 Dec;119(12):2116-2128. doi: 10.1111/add.16581. Epub 2024 Jul 10. PMID 38987890
- [Derived] Collins AB, Baird J, Nimaja E, Ashenafi Y, Clark MA, Beaudoin FL. Experiences of patients at high risk of opioid overdose accessing emergency department and behavioral health interventions: a qualitative analysis in an urban emergency department. BMC Health Serv Res. 2023 Apr 18;23(1):370. doi: 10.1186/s12913-023-09387-7. PMID 37069593
- [Derived] Beaudoin FL, Jacka BP, Li Y, Samuels EA, Hallowell BD, Peachey AM, Newman RA, Daly MM, Langdon KJ, Marshall BDL. Effect of a Peer-Led Behavioral Intervention for Emergency Department Patients at High Risk of Fatal Opioid Overdose: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225582. doi: 10.1001/jamanetworkopen.2022.25582. PMID 35943744
- [Derived] Jacka B, Beaudoin F, Li Y, Nimaja E, Yedinak J, Samuels E, Marshall BDL. Objective Outcome Measures in Randomized Clinical Trials of Interventions to Reduce Risk of Opioid Overdose Following Discharge From the Emergency Department: Utility of Administrative Data Linkage. J Addict Med. 2021 Apr 1;15(2):174-175. doi: 10.1097/ADM.0000000000000705. No abstract available. PMID 32769773
- [Derived] Goedel WC, Marshall BDL, Samuels EA, Brinkman MG, Dettor D, Langdon KJ, Mahoney LA, Merchant RC, Nizami T, O'Toole GA, Ramsey SE, Yedinak JL, Beaudoin FL. Randomised clinical trial of an emergency department-based peer recovery support intervention to increase treatment uptake and reduce recurrent overdose among individuals at high risk for opioid overdose: study protocol for the navigator trial. BMJ Open. 2019 Nov 11;9(11):e032052. doi: 10.1136/bmjopen-2019-032052. PMID 31719087